CLINICAL TRIAL: NCT04933721
Title: An Open-label Study to Provide Berotralstat Access to Subjects With Type 1 and 2 Hereditary Angioedema Who Were Previously Enrolled in Berotralstat Studies
Brief Title: Open-label Berotralstat Access to HAE Patients Previously Enrolled in Berotralstat Studies
Acronym: APeX-A
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BCX7353-312
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Angioedema; HAE
Keywords: prophylaxis
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat

STUDY DESIGN:
Intervention Model Description: Open-label berotralstat (BCX7353) orally administered QD.
Masking Description: No masking as this is open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BCX7353 capsules or granules once daily (Experimental): Berotralstat (BCX7353) capsules or granules orally administered once daily.
  Interventions: Drug: berotralstat

INTERVENTIONS:
Drug: berotralstat — BCX7353 capsules or granules administered orally once daily
  Other Names: Orladeyo

SUMMARY:
This is a phase 3b open-label study providing access to berotralstat for HAE patients who were previously enrolled in berotralstat studies.

DETAILED DESCRIPTION:
APeX-A, 7353-312, is a single-arm, open-label, multicenter study. The study will be conducted in countries where berotralstat is not available either commercially or via another mechanism and is planned in countries where pediatric participants have been enrolled in BCX7353-304 (Study 304). Adult and adolescent (≥12 years) participants will receive berotralstat 150 mg administered orally once daily (QD). Pediatric participants will receive a weight-appropriate dose. The study will assess the long term safety and tolerability of berotralstat.

Eligible subjects will be enrolled directly into Study BCX7353-312 (Study 312) from Studies 302, 204, and 304. Subjects will receive berotralstat administered orally once daily (QD). Subjects will return to the clinic every 24 weeks for drug dispensation and safety monitoring. Participants form Studies 302 and 204 may remain on study for up to 480 weeks (approximately 10 years). Participants from Study 304 may remain in the study until 16 years of age and have access to berotralstat via another mechanism; or up to 5 years, whichever comes first.

Safety and tolerability will be evaluated through assessment of serious adverse events (SAEs) and treatment-related, treatment-emergent adverse events (TEAEs). Up to 139 subjects are planned to enroll.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females currently enrolled in BioCryst-sponsored Study 302, 204, or 304
* Participant or parent/legally designated representative (for participants <18 years of age) able to provide written informed consent.
* Would benefit from continued berotralstat treatment
* Acceptable effective contraception

Key Exclusion Criteria:

* Pregnancy or breast-feeding
* Any condition or situation, including medical history that, in the opinion of the investigator or sponsor, would interfere with the subject's safety or ability to participate in the study
* Use of other medications for long-term prophylaxis of HAE attacks at the Baseline visit or any time during the study.
* Use of any other investigational medicinal product at the Baseline visit or any time during the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2031-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of subjects with a treatment-related TEAE | 240 weeks
Number and proportion of subjects who experience a serious adverse event (SAE) | 240 weeks
Number and proportion of subjects who experience a treatment-related Grade 3 or 4 TEAE | 240 weeks
Number and proportion of subjects who experience a treatment-related Grade 3 or 4 treatment-emergent chemistry abnormality | 240 weeks
Number and proportion of subjects who discontinue due to a TEAE | 240 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Grivcheva-Panoska, MD, PhD, Principal Investigator — PHI University Clinic of Dermatology
Locations (16):
- Study Center, Ottawa, Canada
- Czechia (2):
  - Study Center, Brno
  - Study Center, Pilsen
- France (3):
  - Study Center, Grenoble
  - Study Center, Marseille
  - Study Center, Paris
- Study Center, Frankfurt, Germany
- Study Center, Skopje, North Macedonia
- Study Center, Krakow, Poland
- Study Center, Martin, Slovakia
- Study Center, Cape Town, South Africa
- South Korea (3):
  - Study Center, Daegu
  - Study Center, Gwangju
  - Study Center, Seoul
- Study Center, Madrid, Spain
- Study Center, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No